CLINICAL TRIAL: NCT00640861
Title: MUC1/HER-2/Neu Peptide Based Immunotherapeutic Vaccines for Breast Adenocarcinomas
Brief Title: Vaccine Therapy in Treating Patients With Previously Treated Stage II or Stage III Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000589446; P30CA015083 (NIH); MC0338 (Other: Mayo Clinic Cancer Center); NCI-2009-01342 (Registry Identifier: NCI-CTRP); 782-05 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-03-20; First posted 2008-03-21 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IA breast cancer; stage IB breast cancer; triple-negative breast cancer; HER2-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — CPG-oligonucleotide; incomplete Freund's adjuvant; sargramostim; Immunoenzyme Techniques; Immunologic Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: CpG oligodeoxynucleotide
Biological: HER-2/neu peptide vaccine
Biological: MUC-1 peptide vaccine
Biological: incomplete Freund's adjuvant
Biological: sargramostim
Other: immunoenzyme technique
Other: immunologic technique

SUMMARY:
RATIONALE: Vaccines made from peptides may help the body build an effective immune response to kill tumor cells. It is not yet known which vaccine is most effective in treating breast cancer.

PURPOSE: This randomized clinical trial is studying the side effects of three different vaccine therapies and comparing the vaccines to see how well they work in treating patients with previously treated stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the safety and immunization efficacy of MUC1 and HER-2/neu peptide vaccines combined with CpG oligodeoxynucleotide, sargramostim (GM-CSF), or both, as immune adjuvants suspended in Freund's incomplete adjuvant in patients with previously treated stage II or III adenocarcinoma of the breast.

Secondary

* To describe the impact of immunization on clinical outcomes in patients with MUC1-positive breast cancer in terms of disease-free survival and overall survival.

OUTLINE: Patients are stratified according to Her-2/neu status (positive vs negative). Patients are randomized to 1 of 3 treatment arms.

* Arm A: Patients receive a vaccine comprising incomplete Freund's adjuvant, MUC1 antigen vaccine, two Her-2/neu peptide-based vaccines, and sargramostim (GM-CSF) subcutaneously (SC) on day 1.
* Arm B: Patients receive a vaccine comprising incomplete Freund's adjuvant, MUC1 antigen vaccine, two Her-2/neu peptide-based vaccines (one of them different than in arm A), and CpG oligodeoxynucleotide SC on day 1.
* Arm C: Patients receive a vaccine comprising incomplete Freund's adjuvant, MUC1 antigen vaccine, two Her-2/neu peptide-based vaccines (one of them different than in arm A; the same as in arm B), GM-CSF, and CpG oligodeoxynucleotide SC on day 1.

In all arms, treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients who complete 6 courses of treatment without disease recurrence or a second primary or intolerable toxicity will go to the observation phase of the study for up to 2 years. Patients who develop recurrent disease during the observational phase will go to the event monitoring phase for up to 2 years.

Blood samples are collected periodically. Blood samples and tissue samples from the patient's most recent surgery are used for correlative studies including immune responses to T helper and CTL epitopes by Elispot and tetramer analysis; and antigenic profiling by expression analysis of class I HLA antigens, MUC1, and HER-2 in tumor tissue.

After completion of study treatment, patients are followed periodically until disease recurrence or for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * Clinical stage II or III disease
  * No radiographic evidence of disease at the time of enrollment
  * Has undergone surgery, adjuvant chemotherapy, and/or radiotherapy

    * Completed "standard first-line therapy" only (including adjuvant therapy) for breast cancer within the past 3 months and currently with no evidence of disease
  * Patients with stage I breast cancer with high-risk features are eligible provided 1 of the following criteria are met:

    * HER2 over-expression or amplification
    * Triple-negative (i.e., no expression of ER, PR, or over-expression of HER2 on routine immunohistochemical staining)
* .
* MUC1-positive breast cancer
* HLA-A2 positive
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status 0-2
* Hemoglobin ≥ 8.0 g/dL
* Platelet count ≥ 75,000/μL
* ANC ≥ 1,500/uL
* Creatinine ≤ 2 times upper limit of normal (ULN)
* AST ≤ 2 times ULN
* No uncontrolled infection
* No known HIV infection
* No other circumstances (e.g., concurrent use of systemic immunosuppressants or immunocompromising condition) that in the opinion of the physician would render the patient a poor candidate for this trial
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior invasive malignancies within the past 5 years (with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Fully recovered from acute, reversible effects of any prior breast cancer therapy
* No more than 3 years since prior surgery for primary breast cancer
* Concurrent anti-estrogen therapy is allowed
* No other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-FDA-approved indication and in the context of a research investigation)
* No concurrent enrollment in any other study involving a pharmacologic agent (drugs, biologics, immunotherapy approaches, gene therapy) whether for symptom control or therapeutic intent

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2008-08-28 (Actual); Primary Completion 2015-04-21 (Actual); Study Completion 2015-04-21 (Actual)

PRIMARY OUTCOMES:
Percentage of CD4+ T cells, CD8+ T cells, B cells, monocytes, and dendritic cells in a patient's peripheral blood sample as estimated by flow cytometry with a panel of monoclonal antibodies
Frequency of peptide-specific IFN-gamma producing T cells and peptide-specific IL-5 producing T cells estimated by ELISPOT after in vitro stimulation with peptide-sensitized stimulator cells for MUC1 and HER-2 peptides
Number and severity of hematologic and non-hematologic toxicities reported using the NCI-CTC version 3.0 criteria

SECONDARY OUTCOMES:
Disease-free survival, defined as the time from registration to the documentation of a first failure where a failure is the recurrence of breast cancer or a diagnosis of a second primary cancer
Overall survival, defined as the time from registration to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir Markovic, MD, PhD, Study Chair — Mayo Clinic; Barbara A Pockai, M.D., Principal Investigator — Mayo Clinic; Edith A Perez, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota